CLINICAL TRIAL: NCT05191641
Title: Evaluation of the Effect of Individualized Nursing Care Based on the Professional Values Model for Parents of Pediatric Oncology Patients: A Randomized Controlled Trial
Brief Title: Effect of Individualized Nursing Care for Parents of Pediatric Oncology Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ayla Kaya, Research Assistant Dr., Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AkdnzUnvrsty
Record Dates: First submitted 2021-12-03; First posted 2022-01-13 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Parents; Oncology
Keywords: child; parent; oncology; nurse; education; model
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Single-blind randomized controlled study
Who Masked: Outcomes Assessor
Masking Description: The statistician will be blind in evaluating the results. The intervention and control group will be defined as group 1 and group 2 for statistical analysis. Scales will be evaluated by the researcher who cannot be blinded due to the nature of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (Experimental): PVQ and PedsQL will be used to collect research data. The same measurement tools will be used in the collection of pre-test, mid-term and post-test data. After obtaining the necessary written and verbal permissions from the parents in the intervention group included in the research, 12-week individualized nursing care will be applied. It is planned to make three measurements, namely pre-test, interim evaluation and post-test, from the parents in the intervention groups.
  12 Weeks of Individualized Nursing Care
  * 5 individual interviews
  * A interview after 2 weeks
  * Telephone consultation
  Interventions: Other: Individualized nursing care
- Control group (No Intervention): Pre-test (PVQ and PedsQL) will be applied after obtaining informed consent from the parents included in the control group after randomization. In the pre-test application, an interim evaluation (PVQ and PedsQL) will be applied to the control group 1 week after and the post-test (PVQ and PedsQL) will be applied 4 weeks later. After the post-test application is completed, a five-day individual interview will be applied to the parents included in the control group.

INTERVENTIONS:
Other: Individualized nursing care — Individualized nursing care based on the Professional Values Model for parents of pediatric oncology patients
  Arms: İntervention group

SUMMARY:
Objective: This study was planned to evaluate the effectiveness of individualized nursing care based on the Professional Values Model for parents of pediatric oncology patients.

Method: Simple randomization will be used to evaluate the intervention and control groups. The sample of the study will be the parents of children aged 1-18 years (Intervention group: 35 parents, Control group: 35 parents) diagnosed with cancer in the Akdeniz University Hospital Pediatrics, Hematology and Oncology clinic and hospitalized. Portrait Values Questionnaire and PedsQL Health Care Satisfaction Hematology/Oncology Module Parent Form will be used to collect data. A 12-week individualized nursing care based on the Professional Values Model will be applied to 35 parents in the intervention group. The effectiveness of the program will be evaluated after all post-test applications are completed.

DETAILED DESCRIPTION:
Study Design: A single-blind, randomized controlled trial

Participants and Setting: The population of the research will be the parents of the children hospitalized in the Pediatrics, Hematology and Oncology Clinic of Akdeniz University Hospital. Parents who agreed to participate in the research (Intervention group: 35 parents, Control group: 35 parents) will form the sample of the research. Simple randomization will be used to evaluate the intervention and control groups.

Randomization, allocation, and blinding: After obtaining informed consent from the parents, each will be given a unique sequence number in a sealed envelope. In this study, random selection of participants and assignment to groups will be done by a nurse at the clinic where the research was conducted. Thus, the researcher who implements the training will be blinded. The Consolidated Reporting Standards (CONSORT) flowchart (Moher et al., 2012) will be followed to manage the random allocation process. The 12-week individualized nursing care practice will be carried out by a nurse with sufficient communication skills, 11 years of pediatric oncology clinical and responsible nursing experience, and a doctoral degree in pediatric nursing in the study team. Thus, the difference that may arise from the educator will be eliminated. Depending on the nature of the intervention administered, researchers and participants will not be blinded. The data will be analyzed by the statistician who is unaware of the intervention and control groups. Thus, it will be possible to be blind in terms of statistics and reporting.

Instruments: Parent Descriptive Information Form, Portrait Values Questionnaire (PVQ) and Pediatric Quality of Life Inventory (PedsQL) Health Care Satisfaction Hematology/Oncology Module Parents Form will be used to collect data. Parent Descriptive Information Form was created by the researchers in order to determine the socio-demographic characteristics of the sample. Form consists of a total of 15 items. PVQ is a 40-item scale developed by Schwartz et al. (2001) to measure individuals' value orientations more effectively. Participants were asked to mark how similar the items were to themselves with a 6-level rating. The scale consists of 40 items and 10 sub-dimensions. The sub-dimensions are described as follows. Turkish validity and reliability was established (Demirutku & Sümer, 2010). PedsQL was developed by James Varni et al. in 2000 and adapted into Turkish in 2012 by Kürtüncü Tanır and Kuğuoğlu. PedsQL; 1) general satisfaction (3 items), 2) knowledge (5 items), 3) family involvement (4 items), 4) communication (5 items), 5) technical skills (4 items), 6) emotional needs (4 items) It is a versatile inventory consisting of 25 items. The inventory has only the parent form. In the inventory prepared according to the five-point Likert system, it is expressed as I am not satisfied (1), I am not satisfied (2), I am undecided (3), I am satisfied (4) and I am very satisfied (5).

Data collection: The data will be collected in a time period that will not disrupt the care practices of the sick child, at the place and time deemed appropriate by the clinical nurse and the parent.

İntervention Group The research will be implemented in five stages.

Stage 1: Obtaining the permission of the ethics committee and the institution related to the research

Stage 2: Preliminary Application of the Research. - Preliminary practice will be conducted with the parents of five children hospitalized in the clinic in order to evaluate the intelligibility and applicability of the individualized nursing care content developed on the basis of the Professional Values Model. Parents included in the preliminary application will not be included in the research sample.

Stage 3: Implementation

* Pre-test (PVQ and PedsQL) will be applied after obtaining informed consent from the parents included in the intervention group after randomization.
* Individual interviews will be held for five days, one meeting each day, with the parents included in the initiative group. The contact information of the research team will be shared with the parent.
* During the five-day individual interviews, the knowledge, skills and training needs of the parents and counseling support will be provided by the research team.
* After a five-day individual interview, a break-in interview will be held two weeks later, questions will be answered, and the parent will be counseled over the phone in a 12-week period.

Stage 4: Interim Evaluation

- Interim evaluation (PVQ and PedsQL) will be made 1 week after the pre-test application.

Stage 5: Post-Testing and Evaluation

* The post-test (PVQ and PedsQL) will be applied 4 weeks after the end of the five-day individual interview.
* After the final test data collection phase of the research is completed, the data obtained will be analyzed using the Statistical Package of Social Science (SPSS) 23.0 software package program. The process of evaluating the data will be carried out with the support of a statistician.

Professional Values Model

The Professional Values Model (PDM), which will guide this study, was developed by Kaya and Boz (2019). This model has the feature of being the first theoretical model developed for nurses in Turkey. The framework of the model consists of three basic concepts: "Individual Values", "Professional Values of Nurses" and "Quality of Nursing Care". In the model, the logical relationship between these basic concepts is explained and the importance of individual and professional values, patient satisfaction and increasing the job satisfaction of nurses, as a result, responsibilities in reaching quality nursing care are defined. According to the assumption in the model; the effort to increase the individual values of the individuals receiving care increases the satisfaction of nursing care and the quality of nursing care. Based on this assumption in the model, the nursing care to be applied in this study was developed on the basis of the Professional Values Model.

Individual Interviews Regarding Parents' Care Needs

Interview 1

First meeting, intimate communication with the parent Explanation of the purpose and importance of the study and pre-test application Parents sharing their individual characteristics and experiences, Encouraging the parent to ask questions, determining the need for care in the next meeting

Interview 2

Elimination of the priority maintenance requirement identified in the previous session Determining the parent's perception of health and illness and discussing it on the subject Encourage parents to ask questions and express themselves Determining the maintenance need to be eliminated at the next meeting

Interview 3

Elimination of the priority maintenance requirement identified in the previous session Allowing parents to share their difficulties, experiences, and feelings Enabling the parent to communicate with other patients in the clinic Determining the maintenance need to be eliminated at the next meeting

Interview 4

Elimination of the priority maintenance requirement identified in the previous session Discussion of solutions for the solution of the problems experienced with the parents, the methods used in coping and support systems, and counseling Identifying parental concerns and providing counseling Determining the maintenance need to be eliminated at the next meeting

Interview 5

Elimination of the priority maintenance requirement identified in the previous session Arrangement of the parent's clinic room in accordance with the needs of the curative care environment Post-test application and sharing contact information with the child and parent, informing that they can communicate at any time if needed.

Control Group

* Pre-test (PVQ and PedsQL) will be applied after obtaining informed consent from the parents included in the control group after randomization.
* In the pre-test application, an interim evaluation (PVQ and PedsQL) will be applied to the control group 1 week after and the post-test (PVQ and PedsQL) will be applied 4 weeks later.
* After the post-test application is completed, a five-day individual interview will be applied to the parents included in the control group.

Measurement and Evaluation:

Portrait Values Questionnaire and Pediatric Quality of Life Inventory Health Care Satisfaction Hematology/Oncology Module Parents Form will be used to collect research data. The same measurement tools will be used in the collection of pre-test, mid-term and post-test data. After obtaining the necessary written and verbal permissions from the parents in the intervention group included in the research, 12-week individualized nursing care will be applied. No intervention will be applied to the control group. It is planned to make three measurements, namely pre-test, interim evaluation and post-test, from the parents in the intervention and control groups. After the final test data collection phase of the research is completed, the data obtained will be analyzed using the Statistical Package of Social Science (SPSS) 23.0 software package program. The process of evaluating the data will be carried out with the support of a statistician.

Ethical Considerations

Approval from the Akdeniz University Ethics Committee and the necessary written permissions from the Akdeniz University Hospital, where the research will be conducted, will be obtained in order to conduct the research. During individual interviews, the duration of the meeting will be kept as short as possible and the distance between people will be at least 1.5 meters (preferably 2 meters). Everyone in the room will wear a mask during their stay. The windows will be opened and the room will be ventilated frequently. Before starting the study, when the parents are first met, clear and understandable information about the aims of the research and the steps to be followed will be presented by the researcher. It will be made clear that participation in the study is voluntary and that refusal to participate will not affect the care received in the clinic. Before the application of the research, the parent will be informed verbally or in writing about the research and informed consent will be obtained. After the post-test application is completed, the five-day individual interview will also be applied to the parents included in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Being the parent of a pediatric oncology patient
* Speak and understand Turkish

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-09-14 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Individual values awareness level | Individual values awareness level of parent will be evaluated 3 times: pre-test, 1 week after the pre-test, and 12 weeks after the pre-test. The increase in both the mid-term and post-test scores in the 12-week period is the outcome measure.
  An increase in parents' awareness of their individual values is a measure of outcome. This increase will be measured by the "Portrait Values Questionnaire". The higher the average score, the higher the awareness of individual values. Statistical significance will be set at p < 0.05. One week after the "pre-test" for the intervention group, an "intermediate evaluation" will be made with the same measurement tool. In the interim evaluation, it will be evaluated whether there is an increase according to the pre-test score. 12 weeks after the "Portrait Values Questionnaire" and the "pretest", the same group will be given a "posttest" with the same measurement tool. In the post-test, it will be evaluated whether there is an increase in the mid-test and pre-test scores. If there is an increase in both "interim evaluation" and "post-test" scores compared to the "pretest" scores, it can be stated that the training program is effective on individual values.
Parent satisfaction level | Parent satisfaction level will be evaluated 3 times: pre-test, 1 week after the pre-test, and 12 weeks after the pre-test. The increase in both the mid-term and post-test scores in the 12-week period is the outcome measure.
  The increase in the level of awareness of the satisfaction level of the parents is a measure of outcome. This increase will be measured by the "Pediatric Quality of Life Inventory Health Care Satisfaction Hematology/Oncology Module Parents Form". The higher the average score, the higher the parent satisfaction. Statistical significance will be set at p < 0.05. One week after the "pre-test" for the intervention group, an "intermediate evaluation" will be made with the same measurement tool. In the interim evaluation, it will be evaluated whether there is an increase according to the pre-test score. 12 weeks after the "pretest", the same group will be given a "posttest". In the post-test, it will be evaluated whether there is an increase in the mid-test and pre-test scores. If there is an increase in both "interim evaluation" and "post-test" scores compared to the "pretest" scores, it can be stated that the training program is effective on parent satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ayla Kaya, PhD, Study Director — Akdeniz University Faculty of Nursing
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaya A, Boz I. The development of the Professional Values Model in Nursing. Nurs Ethics. 2019 May;26(3):914-923. doi: 10.1177/0969733017730685. Epub 2017 Sep 20. PMID 28929939
- [Background] • Demirutku, K. Sümer, N. Temel değerlerin ölçümü: portre değerler anketinin türkçe uyarlaması. Türk Psikoloji Yazıları, 2010; 13(25), 17-25
- [Background] • Kürtüncü Tanır M, Kuğuoğlu S. Pediatrik Yaşam Kalitesi Envanteri (PedsQL) Sağlık Bakım Memnuniyeti Hematoloji/Onkoloji Modülü Ebeveyn Formu Geçerlik-Güvenirliliği. Ankara Sağlık Hizmetleri Dergisi, 2012; 11(2).
- [Background] Pai AL, Greenley RN, Lewandowski A, Drotar D, Youngstrom E, Peterson CC. A meta-analytic review of the influence of pediatric cancer on parent and family functioning. J Fam Psychol. 2007 Sep;21(3):407-15. doi: 10.1037/0893-3200.21.3.407. PMID 17874926
- [Background] • Schwartz, S. H., Melech, G., Lehmann, A., Burgess, S., Harris, M. ve Owens, V. (2001). Extending the cross-cultural validity of the theory of basic human values with a different method of measurement. Journal of Cross- Cultural Psychology, 32, 519-542.
- [Background] Harper FW, Peterson AM, Albrecht TL, Taub JW, Phipps S, Penner LA. Satisfaction with support versus size of network: differential effects of social support on psychological distress in parents of pediatric cancer patients. Psychooncology. 2016 May;25(5):551-8. doi: 10.1002/pon.3863. Epub 2015 Jun 17. PMID 27092714
- [Background] Çiftcioğlu, Ş., & Efe, E. (2017). Validity and Reliability of the Oral Assessment Guide for Children and Young People Receiving Chemotherapy. Turkish Journal of Oncology/Türk Onkoloji Dergisi, 32(4).